CLINICAL TRIAL: NCT06907485
Title: A Multicenter Study to Assess the Feasibility of Gleolan (ALA / Aminolevulinic Acid HCl) in Pediatric Brain Tumor Patients After Delayed Administration
Brief Title: A Multicenter Study to Assess the Feasibility of 5-Aminolevulinic Acid (5-ALA) in Pediatric Brain Tumor Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Costas Hadjipanayis (Other)
Collaborators: NX Development Corp (Industry); Southeastern Brain Tumor Foundation (Unknown); StacheStrong Foundation (Unknown); Neuroscience Research Foundation (Unknown); University of Pittsburgh Medical Center (Other); Advocate Hospital System (Other)
Responsible Party: Sponsor-Investigator, Costas Hadjipanayis, L. Dade Lunsford Professor of Neurosurgery, Executive Vice Chairman, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY22120058
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Brain Tumor
Keywords: Aminolevulinic Acid (ALA); Gleolan®; Fluorescence-Guided Resection; Brain Tumor; Pediatric
MeSH Terms: conditions — Brain Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aminolevulinic acid hydrochloride (Experimental): Single arm study administering a single oral solution of aminolevulinic acid hydrochloride at a dose of 20 mg/kg body weight, 6-12 hours prior to brain surgery for resection of the tumor.
  Interventions: Drug: Aminolevulinic acid hydrochloride

INTERVENTIONS:
Drug: Aminolevulinic acid hydrochloride — Pediatric patients diagnosed with a new or recurrent brain tumor, suspected to be either a high-grade or low-grade glioma, and scheduled for surgical removal will receive aminolevulinic acid hydrochloride prior to surgery for resection of the brain tumor.
  Other Names: Gleolan®; ALA HCl; 5-ALA; Aminolevulinic acid HCl; Aminolevulinic acid

SUMMARY:
This clinical trial focuses on pediatric patients aged 2 up to 18 years of age with a new or recurrent pediatric brain tumor, suspected to be either a high-grade or low-grade glioma, and scheduled for surgical removal. 5-aminolevulinic acid (5-ALA) is FDA-approved for improving brain tumor visualization in adults during surgery through fluorescence, enabling more complete removal of the tumor. This study aims to evaluate the feasibility of administering 5-ALA to pediatric brain tumor patients and to assess the quality of tumor fluorescence during surgery in this patient population.

For the clinical trial, the patient will orally ingest 5-ALA 6 to 12 hours before brain surgery. All study participants will be provided standard medical care for removal of the brain tumor. All children enrolled in the study will be closely monitored prior to, during, and after surgery to ensure there are no reactions to the study drug. 5-ALA can make the patient more sensitive to sunlight and direct indoor lighting, referred to as photosensitivity, and can cause a sunburn-type reaction. It is for this reason that patients will be kept in subdued light conditions for 48 hours following surgery. Study participation starts once the patient is enrolled in the study until 6-month post-surgery.

DETAILED DESCRIPTION:
The aim of this study is to assess the feasibility of administering 5-ALA pre-operatively and to access if the resulting 5-ALA-induced tumor fluorescence is adequate for fluorescence-guided brain tumor resection in pediatric patients.

In this single-arm, multicenter study, the guardians of the pediatric patient with a newly diagnosed or select recurrent brain tumors will provide consent for the administration of 5-ALA. In relevant cases, assent from the pediatric patients will also be obtained. A total of twenty pediatric brain tumor patients will be treated to evaluate the feasibility of using 5-ALA in this population. All enrolled patients will receive an oral solution of 5-ALA at a dose of 20mg/kg body weight 6-12 hours prior to surgery, followed by tumor resection using either the institutional standard of care or the surgeon's preferred technique.

Resection of fluorescent and non-fluorescent areas will proceed at the surgeon's discretion and the surgeon will indicate the fluorescence of each section. The fluorescence will be characterized as 'none', 'weak,' 'moderate,' or 'strong'; and described as 'patchy' or 'uniform'. When positive fluorescence is present, fluorescence-guided surgery will be performed under white light visualization with the ability to select for the use of appropriate filters adapted to the surgical microscope to allow specific wavelength of blue light to excite the tumor tissue during the operative procedure. Tissue fluorescence will be recorded by intraoperative photography. Biopsies, routinely performed during surgical tumor resection, will be obtained. An additional three to six research tissue specimens will be collected per patient for histopathologic analysis. If fluorescence is present in the tumor, three fluorescent specimens will be obtained from the tumor-core, tumor-margin, and regions just distant to the tumor margins as well as three non-fluorescent tissue specimens will be obtained adjacent to the resection cavity. If no fluorescence is visualized, this will be documented, and only three samples of non-fluorescent tissue specimens will be obtained from the tumor-core, tumor-margin, and regions just distant to the tumor margins.

Histopathologic analysis on all collected fluorescent and non-fluorescent tissue specimens will be performed by a neuropathologist who will not be informed of the fluorescence status of the tissue specimens. The neuropathologist will characterize the biopsies and the additional three to six research tissue specimens by WHO grade, tumor type, and the number of tumor cells present. If institutions perform routine genetic and molecular analysis on resected tissue, this data will also be collected.

5-ALA makes a person more sensitive to sunlight and direct indoor lighting, referred to as photosensitivity, and can cause a sunburn-type reaction. Skin photosensitization lasts from approximately 24 to 48 hours following 5-ALA administration. It is for this reason that patients will be kept in low light conditions for 48 hours following surgery.

Patients will undergo standard of care clinical assessments, including physical exams, neurological assessments (Karnofsky Performance Scale and the Lansky Scale), and laboratory evaluations, at several time points: upon entry into the trial (before surgery), within 48 hours after surgery, 2-weeks post-surgery, 6-weeks post-surgery, 3-months post-surgery, and 6-months post-surgery. MRIs will be conducted as part of standard care before surgery, within 48 hours of surgery, and at 3-months post-surgery, and 6-months post-surgery. All patients enrolled on the study will be monitored according to the protocol for 6-months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects included in this trial must have had an MRI documentation of "a new or recurrent primary pediatric brain tumor" for which resection is indicated and has been planned.
2. The anticipated histology at resection will be "newly diagnosed" or "recurrent": pilocytic astrocytoma, pleomorphic xanthoastrocytoma (PXA), ganglioglioma, diffuse neuroepithelial tumor (DNET), astrocytoma, oligodendroglioma, ependymoma, anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic ependymoma, anaplastic ganglioglioma, anaplastic PXA, PNET, ATRT, or medulloblastoma.
3. Male or Female Age 2-17 years and 182 days
4. Subjects must have normal organ and marrow function as defined below:

   Leukocytes >3,000/mL Platelets >100,000/mL Total bilirubin Below upper limit of normal (ULN) AST (SGOT)/ALT (SGPT)/ GGT <2.5 X institutional age-specific ULN Creatinine Below ULN

   OR

   Creatinine Clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional age-specific normal as defined per institution.
5. The effects of 5-ALA on the developing human fetus are unknown. A pregnancy test will be performed for all young women of childbearing ability prior to surgery (see Exclusion Criteria below). Should a young woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
6. Ability for patient/patient's guardian to understand and the willingness to sign a written informed consent document. In appropriate cases, assent of pediatric patients will be obtained. Translation will be provided as appropriate.
7. Inclusion of Women and Minorities: Both males and females and members of all ethnic groups are eligible for this trial.

Exclusion Criteria:

1. Patients who meet inclusion criteria but are unable to swallow 5-ALA solution.
2. Patients with radiographic tumors of the brain stem as assessed by MRI.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to 5-ALA. Patients should refrain from use of other potential phototoxic substances (e.g., tetracyclines, sulfonamides, fluoroquinolones, hypericin extracts) for 24 h.
4. Personal or family history of porphyria.
5. Uncontrolled concurrent illness including, but not limited to: ongoing or active infection, heart disease, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with 5-ALA breastfeeding should be discontinued if the mother is treated 5-ALA.
6. Young women who are pregnant or become pregnant will be excluded from the trial as it is unknown if 5-ALA is teratogenic or has abortifacient effects. A pregnancy test will be performed on all young women who are s/p menstruation prior to entering study.
7. Prior history of GI perforation, diverticulitis, and/or peptic ulcer disease.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Overall frequency/rate of positive fluorescence in all patients that receive 5-ALA | Day of Surgery
  Overall frequency/rate of positive fluorescence, which is defined as patients with at least one tissue sample with positive fluorescence (score of at least weak and patchy) after using 5-ALA, in all patients administrated 5-ALA with a suspected primary or recurrent brain tumor that is considered to be a low grade (WHO grade I/II) or high grade (WHO grade III/IV) glioma.

SECONDARY OUTCOMES:
Frequency/rate of positive fluorescence within each tumor type | Day of Surgery
  Presence or absence of fluorescence in each tumor type.
Fluorescence quality in all patients receiving 5-ALA and within each tumor type | Day of Surgery
  Fluorescence will be categorized as 'none,' 'weak,' 'moderate,' or 'strong,' and described as 'patchy' or 'uniform.' If fluorescence is present, surgery will be guided by white light with appropriate filters to excite the tumor tissue. Intraoperative photos will capture tissue fluorescence. Biopsies will be taken, including 3-6 additional research specimens per patient for histopathologic analysis. If fluorescence is present, three fluorescent samples will be collected from the tumor core, margin, and areas near the margin, along with three non-fluorescent samples from the resection cavity. If no fluorescence is seen, only non-fluorescent samples from the tumor core, margin, and surrounding areas will be collected. All samples will undergo histopathological examination by a neuropathologist for WHO grade, tumor type, and cell count. Genetic and molecular analysis data will be collected if available.
Accrual rate for each tumor type | Day of Surgery
  Histopathology assessment will characterize the standard of care biopsies by WHO grade and tumor type. If institutions perform routine genetic and molecular analysis of resected tissue, this data will also be collected.
Determination of the sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of tumor fluorescence. | Day of Surgery
  Sensitivity of 5-ALA induced fluorescence is calculated as proportion of all tumor (confirmed by histopathology analysis) specimens with positive fluorescence. Specificity is the proportion of all tumor (confirmed by histopathology analysis) specimens without the presence of fluorescence. Positive predictive value (PPV) is defined as proportion of tissues with 5-ALA induced fluorescence that were confirmed tumor on histopathology. Negative predictive value (NPV) is the proportion of tissues without fluorescence that were confirmed tumor by histopathology. In addition PPV will also be calculated with the proportion of tissues with no visible 5-ALA-induced fluorescence but with detectable levels of fluorescence through novel detection system that were confirmed malignant on pathology.
Frequency/rate of AE in all patients receiving ALA and for each tumor type | Day of Consent signing, day of surgery; within 48 hours of surgery; 2-weeks post-surgery, 6-weeks post-surgery, 3-months post-surgery, 6-months post-surgery
  All adverse events will be collected from the time of drug administration until 6 months following surgery. In addition, serious adverse events (SAE) will be collected beginning from the time the consent/ assent is obtained. The descriptions and grading scales found in the revised NCI CTCAE version 5.0, which will be utilized for adverse event reporting are available online at http://ctep.cancer.gov/reporting/ctc.html.
6-month progression free survival (PFS) | 6-months post-surgery
  Standard of care, gadolinium-enhanced brain MRI will be obtained at 3- and 6-months after tumor resection to assess surgical field and progression.

CONTACTS AND LOCATIONS:
Overall Officials: Constantinos G. Hadjipanayis, MD, PhD, Study Director — University of Pittsburgh; John Ruge, MD, FAANS, Principal Investigator — Midwest Children's Brain Tumor Center, Advocate Children's Hospital-Park Ridge
Locations (2):
- United States (2):
  - MidWest Children's Brain Tumor Center, Advocate Children's Hospital Park Ridge, Chicago, Illinois
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No